CLINICAL TRIAL: NCT03603314
Title: A Two-part, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of SENS-401 in Subjects With Severe or Profound Sudden Sensorineural Hearing Loss
Brief Title: Efficacy of SENS 401 in Subjects With Severe or Profound Sudden Sensorineural Hearing Loss
Acronym: AUDIBLE-S
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SENS 401-201
Record Dates: First submitted 2018-07-05; First posted 2018-07-27 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Severe Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — SENS-401

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 29 mg dose group (Experimental): Patients will receive the study drug (SENS-401) in the form of tablets by mouth, twice a day, during the first 4 weeks after randomization.
  Interventions: Drug: SENS-401
- 43.5 mg dose group (Experimental): Patients will receive the study drug (SENS-401) in the form of tablets by mouth, twice a day, during the first 4 weeks after randomization.
  Interventions: Drug: SENS-401
- placebo oral tablet (Placebo Comparator): Patients will receive the study drug (placebo) in the form of tablets by mouth, twice a day, during the first 4 weeks after randomization.
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: SENS-401 — 29 mg dose group: tablets of 14.5 mg, oral route, by mouth, twice a day, during 4 weeks
  Arms: 29 mg dose group
Other: Placebo Oral Tablet — placebo, oral route, by mouth, twice a day, during 4 weeks
  Arms: placebo oral tablet
Drug: SENS-401 — 43.5 mg dose groupe: tablets of 14.5 mg, oral route, by mouth, twice a day, during 4 weeks
  Arms: 43.5 mg dose group

SUMMARY:
Primary objective of the study is to assess the efficacy of SENS-401 on hearing loss in comparison to placebo at the end of the 4-week treatment period

DETAILED DESCRIPTION:
Patients will receive the study drug (SENS-401 or placebo) in the form of tablets by mouth, twice a day (3 tablets in the morning and 3 tablets in the evening), during the first 4 weeks after randomization.

SENS-401 is an investigational medicinal product. It belongs to a family of drugs known as "5 HT3 antagonist".

ELIGIBILITY:
The main criteria for inclusion:

* Male or female aged at least 18 years old
* Patients with unilateral idiopathic sudden sensorineural hearing loss or unilateral/bilateral acute acoustic trauma leading to sudden sensorineural hearing loss.
* Patients with sudden hearing loss with onset within 96 hours prior to prior to first study drug intake.
* Patients under highly effective contraception

The main criteria for exclusion:

* Bilateral idiopathic hearing loss
* Fluctuating hearing loss
* History of asymmetric hearing (>20 dB difference between ears) to the best knowledge of the patient
* Severe hearing loss (>90 dB) associated with unilateral (ipsilateral) complete vestibular loss.
* History of Ménière's disease, autoimmune hearing loss, radiation-induced hearing loss, acoustic neuroma (schwannoma), otosclerosis, suspected perilymph fistula or membrane rupture, suspected retro-cochlear lesion, or barotrauma
* Previous SSNHL in the affected ear within the past 6 weeks
* Complete loss of peripheral vestibular function on the affected side
* Any drug-based therapy for inner ear hearing loss that is ongoing or was performed in the past 6 weeks (except oral corticosteroids)
* Any ongoing or planned concomitant medication for the treatment of tinnitus until 6 weeks after administration.
* Any therapy known as ototoxic (e.g. aminoglycosides, cisplatin, loop diuretics, quinine etc.) at the current time or in the past 6 months or planned in the coming 3 months.
* Acute or chronic otitis media or otitis externa terminated less than 7 days
* Prior ear surgery of any kind (except ventilating tubes), or cochlear implants
* Known history of, or concomitant severe hepatic, gastrointestinal, cardiovascular, respiratory, neurological (except vertigo or tinnitus), hematological, renal, dermatological or psychiatric disease or substance abuse
* Neurological disorders including stroke, demyelinating disease, brain stem or cerebellar dysfunction within the last 3 months.
* Treatment with any investigational agent within 4 weeks or any past treatment with azasetron or with 5-HT3 antagonists, or any prior or planned treatment by antidepressant treatment containing serotoninergic agents.
* Patients with either a history of significant arrhythmia, or a history of conditions known to increase the proarrhythmic risk (e.g., congestive heart failure, long QT Syndrome, hypokalemia etc...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine HONNET, MD, Study Director — Sensorion
Locations (26):
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Burgas AD Department of Otorhynolaryngology, Burgas
  - MI Minisrty of Interior Affair Sofia Clinic of Otorhinolaryngology, Sofia
  - Military Medical Academy; Clinic of Otorhynolaryngology, Sofia
- Canada (2):
  - CHU de Quebec - Centre Hospitalier de l'Universite Laval, Québec
  - Wall Street ENT Clinic, Saskatoon
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne-Klinika otorinolaryngologie a chirurgie hlavy a krku, Brno
  - Fakultni nemocnice Hradec Kralove -Klinika otorinolaryngologie a chirurgie hlavy a krku, Hradec Králové
- France (7):
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Hôpital Européen, Marseille
  - Hôpital Lariboisière, Paris
  - 109ème Antenne Médicale de Saint-Maixent l'école, Saint-Maixent-l'École
  - 43ème Antenne Médicale de Sarrebourg, Sarrebourg
  - Hôpital d'Instruction des armées SAINTE ANNE, Toulon
  - Hôpital Pierre Paul Riquet- CHU Purpan, Toulouse
- Universitätsklinikum Tübingen Klinik für Hals-, Nasen- u. Ohrenheilkunde Plastische Operationen, Tübingen, Germany
- Israel (4):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Rabin Medical Center, Otolaryngology, Head and Neck Surgery Gour Shasha Tower Building, floor#7, Petah Tikva
- Serbia (2):
  - Clinical Hospital Center Dr Dragisa Misovic-Dedinje, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - MUDr. Igor Kažmér, s.r.o., Liptovský Mikuláš
  - Fakultna nemocnica s poliklinikou J. A. Reimana Presov, Oddelenie otorinolaryngologie a chirurgie hlavy a krku, Prešov
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University Goztepe Training and Research Hospital, Department of Ear,Nose,Throat, Istanbul
  - Erciyes University Medical Faculty Department of Ear Nose Throat, Melikgazi
- The Royal Hallamshire Hospital, Sheffield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Started | 38 | 39 | 38
Completed | 31 | 28 | 35
Not Completed | 7 | 11 | 3
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 3
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet | Total
Number analyzed (Participants) | 38 | 39 | 38 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 36 | 34 | 98
  >=65 years | 10 | 3 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (16.40) | 46.9 (16.01) | 49.8 (14.56) | 50.3 (15.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 9 | 40
  Male | 24 | 22 | 29 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2 | 5 | 2 | 9
  Ethnicity: Not Hispanic or Latino | 36 | 34 | 36 | 106
  Ethnicity: White | NA — Not an ethnicity parameter | NA — Not an ethnicity parameter | NA — Not an ethnicity parameter | NA — Total not calculated because data are not available (NA) in one or more arms.
  Ethnicity: Unknown | NA — Not an ethnicity parameter | NA — Not an ethnicity parameter | NA — Not an ethnicity parameter | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Hispanic or Latino | NA — Not a race parameter | NA — Not a race parameter | NA — Not a race parameter | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Not Hispanic or Latino | NA — Not a race parameter | NA — Not a race parameter | NA — Not a race parameter | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: White | 33 | 31 | 36 | 100
  Race: Unknown | 5 | 8 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Pure Tone Audiometry PTA (dB) (Average of the Hearing Threshold of the 3 Contiguous Most Affected Hearing Frequencies in dB as Identified at Study Entry) From Baseline to the End of Treatment Visit (Day 28 ± 3).
Description: Pure Tone Audiometry PTA (dB) thresholds were determined for each ear at 0.25, 0.5, 1, 2, 3, 4, 6, and 8 kHz for air conduction and 0.5, 1, 2, 3, 4 kHz for bone conduction.
  Pure Tone Audiometry PTA (dB) is an hearing test used to identify hearing threshold levels of an individual and enabling determination of the degree hearing loss.
  A clinically significative improvement is defined as a decrease of at least 10 dB of hearing threshold.
Time Frame: 28 days
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 38 | 39 | 38
dB | -27.754 [-40.534 to -14.974] | -24.931 [-37.793 to -12.069] | -25.214 [-38.310 to -12.119]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; The null and alternative hypotheses for Part 1 of the study were as follows, where μH, μL and μP were defined as the mean change in PTA of the high dose, low dose, and placebo respectively: H0H: μH - μP = 0, HAH: μH - μP <0 (greater decrease on high dose) H0L: μL - μP = 0, HAL: μL - μP <0 (greater decrease on low dose); Test type: Superiority; p = 0.3419, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5181, Mixed Models Analysis

2. Secondary Outcome: Change in Pure Tone Audiometry PTA (dB) (Average of the Hearing Threshold of the 2 Most Affected Hearing Frequencies in dB as Identified at Study Entry) From Baseline to the End of Treatment Visit (Day 28 ± 3).
Description: as for outcome 1
Time Frame: Day 28
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 38 | 39 | 38
dB | -27.910 [-41.211 to -14.610] | -24.468 [-37.860 to -11.076] | -25.726 [-39.369 to -12.084]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3666, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5776, Mixed Models Analysis

3. Secondary Outcome: Change in Pure Tone Audiometry PTA (dB) (the Most Affected Hearing Frequencies in dB as Identified at Study Entry) From Baseline to the End of Treatment Visit (Day 28 ± 3).
Description: as for outcome 1
Time Frame: Day 28
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 38 | 39 | 38
dB | -30.889 [-44.619 to -17.159] | -30.035 [-43.850 to -16.220] | -29.371 [-43.469 to -15.272]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4094, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4602, Mixed Models Analysis

4. Secondary Outcome: Change in Pure Tone Audiometry PTA (dB) (Average of the Hearing Threshold of the 3 Most Affected Hearing Frequencies in dB as Identified at Study Entry) From Baseline to the End of Study Visit (Day 84 ± 3).
Description: as for outcome 1
Time Frame: Day 84
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 33 | 30 | 33
dB | -32.469 [-45.229 to -19.708] | -30.070 [-42.881 to -17.259] | -25.399 [-38.363 to -12.435]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1269, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2257, Mixed Models Analysis

5. Secondary Outcome: Change in Speech Discrimination Threshold From Baseline to Day 28
Description: The Speech recognition threshold (SRT) (dB) is the minimum hearing level at which an individual can correctly recognize 50% of speech material; the more severe the hearing loss is, the higher SRT is. Spondaic words are the usual and recommended test material for the speech recognition threshold; spondaic words are two-syllable words with equal stress on both syllables (eg, birthday). Per the American Speech-Language-Hearing Association (ASHA) guidelines, subjects were familiarized with the spondaic words prior to the test; they listened to the list of words and indicated if any were unfamiliar. These words could then be eliminated from the list.
Time Frame: Day 28
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 38 | 39 | 38
dB | -22.899 [-35.836 to -9.962] | -19.882 [-33.015 to -6.748] | -19.827 [-33.336 to -6.318]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3121, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4965, Mixed Models Analysis

6. Secondary Outcome: Change in Speech Discrimination Threshold From Baseline to Day 84
Description: as for outcome 5
Time Frame: Day 84
Measure: Least Squares Mean (90% Confidence Interval); unit: dB
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
Number analyzed (Participants) | 33 | 30 | 33
dB | -24.990 [-38.040 to -11.940] | -22.671 [-35.939 to -9.403] | -16.642 [-30.236 to -3.048]
Statistical Analysis 1: Comparison: 29 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0976, Mixed Models Analysis
Statistical Analysis 2: Comparison: 43.5 mg Dose Group vs Placebo Oral Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1762, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | 29 mg Dose Group | 43.5 mg Dose Group | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/39 | 1/38
Other Adverse Events (participants affected / at risk) | 20/38 | 13/39 | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 29 mg Dose Group (N=38) | 43.5 mg Dose Group (N=39) | Placebo Oral Tablet (N=38)
diziness (Nervous system disorders) | 0 | 0 | 1 (1)
fatigue (General disorders) | 1 (1) | 0 | 0
headache (Nervous system disorders) | 1 (1) | 0 | 0
colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 29 mg Dose Group (N=38) | 43.5 mg Dose Group (N=39) | Placebo Oral Tablet (N=38)
Constipation (Gastrointestinal disorders) | 10 (11) | 6 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 6 (6) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (5) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT03603314/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03603314/SAP_001.pdf